CLINICAL TRIAL: NCT02007616
Title: Compensation Factors of Cognitive Ageing: Using Computer Technology to Reduce Cognitive Decline in Ageing
Brief Title: Cognitive Aging and Training With Video-games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Principal Investigator, Soledad Ballesteros, Professor Dr., Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSI2010-21609-C02-01
Record Dates: First submitted 2013-12-04; First posted 2013-12-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Aging; Healthy
Keywords: Cognitive aging; Video games training; Attention; Memory; Wellbeing; Speed of processing; Executive functions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-action video game training (Experimental): 20 1-hour sessions of non-action video game training
  Interventions: Other: Non-action video game training
- Control (No Intervention): Participants in the control group did not receive non-action video game training

INTERVENTIONS:
Other: Non-action video game training — Based on cognitive training Lumosity
  Arms: Non-action video game training

SUMMARY:
The ageing of the population will inevitably lead to a growing number of older people living alone and in need of care. Given the high cost of geriatric care, a critical research issue is exploring ways to improve or maintain cognitive and functional status in old age. Unfortunately, it has been shown that training those specific cognitive processes most sensitive to ageing (such as speed of processing or working memory), produces only limited beneficial effects. However, research also suggests that factors such as cognitive engagement, physical activity and social context may act as more general modulators of cognitive decline. This project is a longitudinal study with experimental and control groups. It is inspired from the engagement model of cognitive optimization suggesting that a lifestyle marked by social and intellectual engagement may mitigate age-related declines on cognitive functioning. It uses new cutting-edge information computing technology (ICT) solutions to improve or simply maintain cognitive functions in the elderly. This research investigates how the treatment reduces the effects of cognitive age-related decline in executive control processes and episodic (explicit) memory using behavioral and imaging measures. The results will provide significant knowledge on the potential of new ICT technologies to delay, compensate, and even prevent common chronic problems experienced by the elderly population. The hypothesis is that cognitive training with video-games through ICT solutions will promote brain and mental health and independence. Ultimately, the objective is to contribute to the understanding of factors that help avoiding the (personal and economic) consequences of long-term care in geriatric institutions.

DETAILED DESCRIPTION:
The aim of the present project was to investigate whether older adults could benefit from brain training with video games in a series of cognitive tasks. Two groups of healthy older adults participated in the study. The experimental group received 20 1-hr video game training sessions using a commercially available brain-training package (Lumosity) involving problem solving, mental calculation, working memory and attention tasks. The control group did not practice this package and, instead, attended meetings with the other members of the study several times along the course of the study. Both groups were evaluated before and after the training (experimental group) or a similar period of time (control group) using different cognitive tasks in a 2 (Group: Experimental, control) x 2 (Time os assessment: Pre, post) mixed factorial design.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination (MMSE) score 26 or greater
* Global Deterioration Scale (GDS) score less than 5
* Independent living
* Normal or correct to normal vision and hearing

Exclusion Criteria:

* Diagnosis of dementia
* Planned move from study area
* Inability to complete study activities
* Scores lower than inclusion criteria requirements Communication problems.

Ages: 57 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Neuropsychological testing | Baseline, 12 weeks, and 24 weeks
  Improvement in Neuropsychological tests after training
Oddball task | Baseline, 12 weeks, and 24 weeks
  Improvement in attention after training
Wisconsin task | Baseline, 12 weeks, and 24 weeks
  Improvement in executive functions
Speed of processing task | Baseline, 12 weeks, and 24 weeks
  Improvement in processing speed after training
Spatial working memory (WM) | Baseline, 12 weeks, and 24 weeks
  Improvement in spatial working memory

SECONDARY OUTCOMES:
Efficacy of non-action video game training | Up to 12 weeks
  Efficacy of training: Better performance in the trained video games from first training session to the last training session (from 1 to 20 sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Ballesteros, PhD, Principal Investigator — UNED
Locations (1):
- Facultad de Psicología de la UNED, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Ballesteros S, Mayas J, Prieto A, Toril P, Pita C, Laura Pde L, Reales JM, Waterworth JA. A randomized controlled trial of brain training with non-action video games in older adults: results of the 3-month follow-up. Front Aging Neurosci. 2015 Apr 14;7:45. doi: 10.3389/fnagi.2015.00045. eCollection 2015. PMID 25926790
- [Derived] Mayas J, Parmentier FB, Andres P, Ballesteros S. Plasticity of attentional functions in older adults after non-action video game training: a randomized controlled trial. PLoS One. 2014 Mar 19;9(3):e92269. doi: 10.1371/journal.pone.0092269. eCollection 2014. PMID 24647551
- See also: Web of the Research Group on Studies on Aging and Neurodegenerative Diseases — http://agingandcognitionlab.com/
- See also: Web of the Universidad Nacional de Educación a Distancia — http://portal.uned.es/portal/page?_pageid=93,165833&_dad=portal&_schema=PORTAL
- See also: Lumosity website — http://www.lumosity.com
- See also: PlosOne website — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0092269
- See also: Frontiers website — http://journal.frontiersin.org/Journal/10.3389/fnagi.2014.00277/full